CLINICAL TRIAL: NCT06673420
Title: Enhancing Anatomy Education for First-Year Medical Students Through a Telegram® Channel: a Cross-sectional Study on Learning Augmentation.
Brief Title: Enhancing Anatomy Education for First-Year Medical Students Through a Telegram® Channel
Status: Completed | Type: Observational
Sponsor: Mosab Adam (Other)
Responsible Party: Sponsor-Investigator, Mosab Adam, Principal Investigator, University of Khartoum
Organization: University of Khartoum (Other)
Other Study IDs: NU-REC/11-018/12
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Anatomy Education
Keywords: Anatomy; Telegram; Channel; Medical; Students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- first-year medical students at the University of Khartoum enrolled in the Anatomy thorax module: The total population comprised 360 students. Participation in the Telegram channel created for anatomy learning was voluntary, and the students were given the option to subscribe. No sampling was conducted, to ensure that all students had equal access to the benefits of the channel and we did not wish to exclude anyone ethically. An MCQs test was shared with all students either prescribed or not
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — This is an observational study

SUMMARY:
The goal of this observational study is to evaluate the effects of Telegram channel on anatomy education for fist year medical students and measure students' reflections on it. The main question it aims to answer is: Telegram channel can enhance Anatomy education to the first year medical students.

Participants (either those prescribed or not prescribed to the Telegram channel) answered an online 20-multiple-choice-questions (MCQs) assessment test (summative test).

DETAILED DESCRIPTION:
Ethical Considerations:

Ethical approval for this study was provided by the National University Research Ethics Committee, Khartoum, Sudan on 01/10/2020. The ethical approval number is: NU-REC/11-018/12. All participants consented to participate in the first section of the Google form and written informed consent was obtained from all students who participated in the focus group discussion

Study design and Population:

This prospective cross-sectional study was conducted among first-year medical students at the University of Khartoum enrolled in the thorax module of their Gross Anatomy course. The total population comprised 360 students. Participation in the Telegram channel created for anatomy learning was voluntary, and the students were given the option to subscribe. No sampling was conducted, to ensure that all students had equal access to the benefits of the channel and the investigators did not wish to exclude anyone ethically.

Context and Setting:

The curriculum of Gross Anatomy of Bachelor of Medicine and Surgery at the University of Khartoum is taught over 3 semesters; Thorax and Abdomen in the first semester, Pelvis and Limbs in the second semester, and Head and Neck in the third semester. This study was conducted on first-year medical students enrolled in the thorax module of the undergraduate program, with a total of 360 students. The thorax module is taught for four weeks through dissection room (DR) practical sessions, lectures, and case-based discussions. In the practical sessions, students are divided into small groups each group contains 10 to 12 students and is guided by the practical module through four stations containing prosected cadavers, prosected specimens, plastic models, and dry and plastic bones. Each station is moderated by a departmental tutor. The assessment of the thorax module is performed through a mid-semester exam (which only covers the thorax module) and a final semester exam (which covers both thorax and abdomen modules). Both exams consisted of a spotter test and a written paper test (containing single best-answer questions and short-answer questions).

Telegram Channel:

Telegram allows users to create channels to broadcast messages to large audience members. These channels can have an unlimited number of subscribers who will only receive messages posted by the channel's administration. These messages reach the subscribers directly and appear as notifications on their phones with each post. The channel supports a wide range of content types, from written posts, photos, and auto-playing videos to quizzes and beyond. It also provides the administrators with detailed statistics on the channel's growth and the viewing numbers of its posts. Telegram also allows users to create bots. These are special accounts that can be used to send and receive anonymous messages.

A Telegram channel was created on the 16th of October 2020 under the name "Doses of Human Anatomy". Students were invited to join the channel through an invitation link sent to their cohort's Telegram group. The channel began posting on the 17th of October 2020. It was posting five days a week on a regular basis, from Saturday to Wednesday, over a period of four weeks. These posts were ongoing, in line with the practical sessions of the thorax. On October 29th, a Telegram feedback bot account was created and shared with the channel, allowing students to give feedback about the channel and suggesting specific topics to be targeted by the new posts.

Throughout the one-month study period, quizzes (formative tests different from the summative test, which was done after the end of the thorax module) were created and shared on the channel at the end of every week. These were programmed mini-tests, usually consisting of five questions each. The performance of students ordered by their scores and the time they took to answer the quiz became available to the channel administrators as soon as the answers were submitted. Students also received immediate programmed feedback for any question that they submitted an incorrect answer.

During the study period, the channel posted 17 posts. There were nine written posts with image illustrations, two written posts without image illustrations, five quizzes, and one video.

Assessment, Questionnaire and Focus Group Discussion:

After finishing the thorax module (one month of using the Telegram channel), a Google form containing a 20-multiple-choice-questions (MCQs) assessment test (summative test) and a feedback questionnaire were shared with all students (360 students) on their telegram accounts, telegram groups, and on the telegram channel itself. The questions on the assessment test were set by two independent assessors from the Department of Anatomy at the University of Khartoum. Both assessors were not subscribers to the channel and had no knowledge of the material posted on the channel. The 20 questions covered the entire thoracic module. The feedback questionnaire targeted demographic data, sources of studying anatomy, favorite types of posts, the role of the channel in learning anatomy, and whether students recommend the channel to continue posting or to stop. Sectioning the Google form allowed all first-year medical students in the thorax module to participate in the assessment test, while only subscribers to submit a response the feedback questionnaire.

Focused group discussion:

After the one-week window of receiving responses on the Google form, the form was closed, and the investigators issued a call for students subscribed to the channel to voluntarily participate in a focus group discussion. This call was open for one week, and eight students responded, receiving invitations to participate in the discussion. This FGD was in person and took approximately one and a half hours. Qualitative feedback was collected through six open-ended questions. These questions targeted students' studying approaches, their reflections on the material provided by the channel, the impact of the channel, and their suggestions to improve the channel. The discussion was voice-recorded, and the responses were categorized for further grouping and analysis.

Data Entry and Analysis:

The data was entered automatically from the Google form into an Excel sheet. Data was then analyzed using the Statistical Package for Social Sciences (SPSS) ver22. Descriptive statistics in the form of frequencies, percentages, tables, and figures are presented. Independent sample t-test and Chi-square test were used to assess associations. A p-value was considered significant when less than 0.05 at a confidence level of 95%.

The focus group discussion was recorded, and a Microsoft Word copy of the transcript was created after cleaning and labelling.

ELIGIBILITY:
Inclusion Criteria:

* First Year medical students at the University of Khartoum, Sudan and enrolled in the thorax module of their Gross Anatomy course

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This prospective cross-sectional study was conducted among first-year medical students at the University of Khartoum enrolled in the thorax module of their Gross Anatomy course. The total population comprised 360 students. Participation in the Telegram channel created for anatomy learning was voluntary, and the students were given the option to subscribe. No sampling was conducted, to ensure that all students had equal access to the benefits of the channel and we did not wish to exclude anyone ethically.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
The score of the participants in the summative test | 17/11/2020 to 24/11/2020
  a Google form containing a 20-multiple-choice-questions (MCQs) assessment test which covered the entire thoracic module. The score has a total of 20 points with 0 is the minimum value and 20 is the maximum value. High score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Awad, A. Professor, Study Director — University of Khartoum
Locations (1):
- Anatomy department, University of Khartoum., Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Undecided